CLINICAL TRIAL: NCT01058915
Title: Influence of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on Plaque Composition Assessed by Virtual Histology in Patients With ST-Segment Elevation Acute Myocardial Infarction (VIRHISTAMI)
Brief Title: Influence of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on Plaque Composition in Patients With ST-Segment Elevation Myocardial Infarction (MI)
Acronym: VIRHISTAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Rasmus Egede, Department of Cardiology, Odense University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-003111-43
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Acute Coronary Syndrome
Keywords: ST-Segment Elevation Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin 5mg (Active Comparator): Rosuvastatin 5mg/day for one year
  Interventions: Drug: Rosuvastatin 5mg
- Rosuvaststin 40mg (Active Comparator): Rosuvastatin 40mg/day
  Interventions: Drug: Rosuvastatin 40mg

INTERVENTIONS:
Drug: Rosuvastatin 5mg — Rosuvastatin 5mg/day
  Other Names: Crestor
  Arms: Rosuvastatin 5mg
Drug: Rosuvastatin 40mg — Rosuvastatin 40mg/day
  Other Names: Crestor
  Arms: Rosuvaststin 40mg

SUMMARY:
In patients with ST-segment elevation acute myocardial infarction (STEMI) increased LDL-cholesterol reduction (rosuvastatin 40 mg) will provide incremental plaque stabilization (changes in plaque composition) and plaque regression over 12 months beyond the benefit of moderate LDL-cholesterol reduction (rosuvastatin 5 mg) (assessed by IVUS and VH).

ELIGIBILITY:
Inclusion Criteria:

* ST segment elevation acute myocardial infarction
* 20% < angiographic diameter stenosis < 50% on a not previously revascularized native coronary artery
* Statin naïve

Exclusion Criteria:

* Pharmacologic lipid lowering treatment before index hospitalization
* Atrial fibrillation, not well rate-controlled
* Ventricle frequency variation with more than a factor 2 over 1 minute
* Unconscious patients
* Total cholesterol > 7.0 mmol/l
* History of statin induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins) including rosuvastatin
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception or have a positive serum pregnancy test (a serum-human chorionic gonadotrophin [Beta-HCG] analysis)
* History of malignancy (unless a documented disease free period exceeding 5-years is present) with the exception of basal cell or squamous cell carcinoma of the skin, or in the case of a study designed to investigate antineoplastic properties of rosuvastatin. Women with a history of cervical dysplasia would be permitted to enter the study provided they had 3 consecutive clear Papanicolaou (Pap) smears
* Uncontrolled hypothyroidism (TSH > 1.5xULN)
* Abnormal LFT's
* History of alcohol or drug abuse within the last 5 years (this may affect compliance)
* Current active liver disease (ALT/SGPT >2xULN or severe hepatic impairment (to protect patient safety as directed on the labels of currently approved statins)
* Unexplained creatine kinase (CK > 3xULN) (To protect patient safety) (will be increased at baseline because of acute ST segment elevation myocardial infarction a few days before enrolment)
* Serum creatinine >176mmol/L (2.0mg/dL) (unless the protocol specifically aims to investigate a chronic renal disease population)
* Participation in another investigational drug study less than 4 weeks before enrolment in the study, or according to subjects local ethics committee requirements where a larger period is stipulated (to avoid potential misinterpretation of overlapping adverse events)
* Treatments with cyclosporine
* Treatment with gemfibrozil

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Changes in plaque composition (VH) in a not previously revascularized or infarct related coronary artery with an angiographic insignificant lesion (Follow up - baseline). | One year

SECONDARY OUTCOMES:
Percent changes in plaque volume in a not previously revascularized coronary artery with an angiographic insignificant lesion (Follow up - baseline). | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Egede, MD, Principal Investigator — Department of Cardiology, Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Fuenen, Denmark

REFERENCES:
- [Background] Nair A, Kuban BD, Tuzcu EM, Schoenhagen P, Nissen SE, Vince DG. Coronary plaque classification with intravascular ultrasound radiofrequency data analysis. Circulation. 2002 Oct 22;106(17):2200-6. doi: 10.1161/01.cir.0000035654.18341.5e. PMID 12390948
- [Background] Jensen LO, Thayssen P, Pedersen KE, Stender S, Haghfelt T. Regression of coronary atherosclerosis by simvastatin: a serial intravascular ultrasound study. Circulation. 2004 Jul 20;110(3):265-70. doi: 10.1161/01.CIR.0000135215.75876.41. Epub 2004 Jul 6. PMID 15238460
- [Derived] Egede R, Jensen LO, Hansen HS, Hansen KN, Junker A, Thayssen P. Influence of high-dose lipid lowering treatment compared to low-dose lipid lowering treatment on plaque composition assessed by intravascular ultrasound virtual histology in patients with ST-segment elevation acute myocardial infarction: the VIRHISTAMI trial. EuroIntervention. 2013 Feb 22;8(10):1182-9. doi: 10.4244/EIJV8I10A182. PMID 22987572